CLINICAL TRIAL: NCT04913974
Title: Univation X: A Functional and Clinical Outcomes Study of a Partial Knee Replacement
Brief Title: Univation X Partial Knee Study
Status: Withdrawn | Type: Observational
Why Stopped: Surgeons unhappy with the outcome from pre-study implants
Sponsor: Golden Jubilee National Hospital (Other Government)
Collaborators: Aesculap AG (Industry)
Responsible Party: Sponsor
Other Study IDs: Ortho 17-06
Record Dates: First submitted 2019-07-17; First posted 2021-06-04 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Arthritis
Keywords: unicondylar knee replacement; uni-compartmental knee replacement; knee arthroplasty; gait; motion analysis
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Uni-condylar knee arthroplasty: A cohort of patients who will undergo uni-condylar knee replacement surgery with the Univation X system and have biomechanical anaylsis
  Interventions: Procedure: Uni-condylar knee arthroplasty

INTERVENTIONS:
Procedure: Uni-condylar knee arthroplasty — Surgical replacement of medial compartment of arthritic knee with an implant
  Other Names: uni-condylar knee replacement

SUMMARY:
The objective of this study is to investigate the functional and clinical outcome after medial unicompartmental knee replacement using the Aesculap AG Univation X knee prosthesis compared to pre-operative data and a healthy control group.

DETAILED DESCRIPTION:
All potential medial uni-compartmental knee arthroplasty patients from consultant orthopaedic surgeons at the Golden Jubilee National Hospital (GJNH) will be screened in relation to the inclusion/exclusion criteria. Invitation letters and participant information sheets (PIS) will be sent out to suitable patients who have been referred to the GJNH for a knee replacement (allocated patients) prior to their pre-operative consultation with their surgeon. They will be approached at their consultation visit to seek consent to take part in the study. Patients who have been referred to the GJNH for assessment for a knee replacement (see and treat patients) will be approached only if they are deemed eligible for uni-compartmental knee replacement by their consultant, and will be given a copy of the participant information sheet along with the invitation letter. They will be approached for consent to take part in the study at their pre-operative assessment. All patients will be contacted by telephone around a day after receiving the participant information sheet to ask for verbal consent. This is necessary to arrange the pre-operative CT scans and biomechanical testing. All patients will be given the opportunity to ask questions about the study before signing the consent form. Consent will be taken by the chief investigator or their delegate, using a signed form.

Thirty patients will be recruited to the study. They will have their surgery performed by one of the participating consultants using the study implant, the Univation X unicondylar knee system manufactured by Aesculap AG.

Participants will receive their standard in-patient care and rehabilitation. Standard hospital care for knee arthroplasty patients is for them to return to the hospital for a post-operative review at 6 weeks and then 1 year after operation. Study participants will also be asked to attend the GJNH for one additional research specific appointment at two years post-operatively.

During the standard care appointments, patients will be reviewed by a member of the arthroplasty team who will collect routine data on the clinical and functional outcomes and implant stability. These data include the Oxford Knee Score (OKS), EURO Quality of life questionnaire (EQ-5D 5L), patient satisfaction and standard radiographic assessment of the implant.

Detailed radiographic analysis will be carried out on radiographs collected as standard practice and computed tomography (CT) scans taken specifically for the study. Radiographs will be taken pre-operatively, post-operation at day one (standard), 1 year (standard) and the 2 year (study) time points. Patients will have a CT scan pre-operatively and 6 weeks post-operatively. The post-operative scan will be performed instead of the radiographs usually take at this time point. The pre-operative scan will be performed in addition to the pre-operative radiographs.

Study participants will also have two sessions of specialised functional assessment using clinical movement analysis before surgery and 1 year after surgery during their standard pre- and post-operative visits. Biomechanical movement analysis will be carried out in an on-site movement analysis laboratory. Study participants will be required to wear suitable clothing (e.g. tee shirt and shorts) and be barefoot. A number of reflective markers will be attached to specific locations on the body (using suitable double sided tape) which will be tracked by a number of infrared cameras. Participants will be asked to perform the following tasks; level walking, incline walking, decline walking, stand-to-sit-to-stand, step ascent and descent and single leg balance. Each task will be performed at least three times to enable the collection of three good sets of data. In addition, the two stepping tasks will be repeated for each limb. The single leg balance will be performed once for each leg and data will be collected for 30 seconds per limb. A motion capture system will collect limb and torso movements during the task performances while force plates will collect ground reaction forces.

After the two year follow-up appointment the patients involvement in the study will be complete.

ELIGIBILITY:
Inclusion Criteria:

* Patients having medial uni-compartmental knee arthroplasty Functionally intact anterior cruciate ligament Able to give informed consent Able to return to GJNH for follow-up BMI under 40

Exclusion Criteria:

* Inflammatory joint disease e.g. rheumatoid arthritis Previous hip procedure in the last twelve months Previous knee surgery other than arthroscopy and medial menisectomy Previous ankle surgery Symptomatic foot, hip or spinal pathology Any medical condition limiting normal ambulation e.g. stroke, Charcot-Marie-Tooth disease, severe lymphedema, advanced cardiac disease

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female participants aged between 45 and 75 inclusive under the care of one of the study surgeons who have been listed for uni-condylar knee replacement surgery. They must live locally enough to be intending returning to the hospital for follow-ups rather than opting to be followed-up locally. They should have a BMI of under 40 otherwise skin artifacts would be an issue for the accuracy of the biomechanical analysis. They must have had no previous lower limb arthroplasty in the previous 12 months or conditions which could influence their mobility other than the condition for which they are having arthroplasty for.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-02 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Knee joint angle during step descent | up to 1 year
  Knee angles collected using clinical movement analysis

SECONDARY OUTCOMES:
Oxford Knee Score | Pre-operatively, 6 weeks, 1 year and 2 years post-op
  Patient-reported knee pain and function
EQ5D-5L | Pre-operatively, 6 weeks, 1 year and 2 years post-op
  Patient-reported quality of life
Patient satisfaction | 6 weeks, 1 year and 2 years post-op
  Patient-reported satisfaction of the knee using a five point Likert scale
Implant survivorship | 2 years
  Percentage of implants still in situ over time.
Peri-prosthetic lucency | 6 weeks, 1 year and 2 years post-op
  Radiolucent lines (>2mm wide) around the component which may indicate component loosening
Component position | 6 weeks, 1 year and 2 years post-op
  Migration of the component over time measured from CT scans
Complications | 6 weeks, 1 year and 2 years post-op
  Any post-operative complications as a result of surgery, e.g. infection, revision, aseptic loosening.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Ohly, MBBS, Principal Investigator — Golden Jubilee National Hospital
Locations (1):
- Golden Jubilee National Hospital, Clydebank, West Dunbartonshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No